CLINICAL TRIAL: NCT05854394
Title: Effect of Multimodal Prehabilitation on Functional Recovery and Quality of Life After Colorectal Cancer Surgery
Brief Title: Effect of Multimodal Prehabilitation After Colorectal Cancer Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiamen University (Other)
Responsible Party: Principal Investigator, JiaJun Zhang, Principal Investigator, Xiamen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCT20211154469
Record Dates: First submitted 2023-04-25; First posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Colorectal Cancer
Keywords: Prehabilitation; Quality of life; Cancer-related fatigue; Colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: patients were randomly assigned to the prehabilitation group and control group by online randomization software
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prehabilitation group (Experimental): Multimodal prehabilitation strategy includes physical exercise (moderate aerobic exercise combined with resistance exercise and respiratory training ), nutritional suggestion and optimization#whey protein supplement#, and psychological therapy, as well as conventional guidance (including drug treatment recommendations for chronic disease, quit smoking and abstinence).
  Interventions: Behavioral: Multimodal prehabilitation management Multimodal prehabilitation management
- Control group (No Intervention): The patients will receive the conventional clinical guidance according to The First Affiliated Hospital of Xiamen University, including drug treatment recommendations for chronic disease, quit smoking and abstinence.

INTERVENTIONS:
Behavioral: Multimodal prehabilitation management Multimodal prehabilitation management — Multimodal prehabilitation strategy includes physical exercise (moderate aerobic exercise combined with resistance exercise ), nutritional suggestion and optimization（whey protein supplement）, and psychological therapy, as well as conventional guidance (including drug treatment recommendations for chronic disease, quit smoking and abstinence).
  Arms: Prehabilitation group

SUMMARY:
The process of enhancing an individual's functional capacity to optimize physiologic reserves before an operation to withstand the stress of surgery has been coined prehabilitation. This is a prospective randomized controlled trail, designed to explore if the patients who take Colorectal Cancer Surgery will benefit from short-term multimodal prehabilitation strategy. multimodal prehabilitation includes exercise, nutrition supplement and physiology management preoperatively. It starts from the day that patients decide to take the surgery until the day before surgery, lasting 1~2 week in The First Affiliated Hospital of Xiamen University. And investigators follow-up patients until 4 weeks after surgery to investigate if multimodal prehabilitation strategy can improve the postoperative functional recovery and improve the quality of life #reduce complications and improve prognosis.

DETAILED DESCRIPTION:
The process of enhancing an individual's functional capacity to optimize physiologic reserves before an operation to withstand the stress of surgery has been coined prehabilitation. It has been confirm that trimodal prehabilitation strategy including exercise, diet and psychology guidance could improve postoperative functional recovery after surgery for patients undergoing colorectal resection. Although many clinical studies have confirmed that preoperative exercise for patients undergoing colorectal cancer surgery is safe and useful, but the prehabilitation strategy in previous studies usually takes 4~8 weeks. However, patient suspected of malignant tumor often wouldn't wait for such a long period. Investigators therefore designed this study to investigate if a 1~2 week multimodal prehabilitation strategy benefits the patients undergoing laparoscopic colorectal cancer resection. There will be 100 patients awaiting operation for primary colorectal cancer recruited in this research at The First Affiliated Hospital of Xiamen University.

After informed consent was obtained, the patients will be divided into two groups randomly, the prehibilitation group and control group.

The prehabilitation group will receive an individual trimodal prehabilitation strategy after a complete assessment, including physical exercise, nutritional optimization, and psychological therapy, as well as conventional guidance. The length of prehabilitation was determined by the waiting time till surgery alone. The control group will receive the conventional guidance, including drug treatment recommendations for chronic disease, quit smoking and abstinence. Both of the groups are also provided some useful information about surgery process. The functional capability will be examined for both groups at several time points (baseline, the day before surgery,4 weeks postoperatively) The primary end point is functional walking capacity as measured by the 6 minutes walking distance (6MWD) 4 weeks postoperatively, health-related quality of life scales and cancer-related fatigue. The secondary end points include self-reported physical activity, and prognosis information (postoperative complications, length of hospital stay, ICU stay time, hospitalization expenses, etc.).

ELIGIBILITY:
Inclusion Criteria:

* From 18 y/o to 75 y/o
* Suspected of colorectal cancer
* Decide to take the colorectal cancer radical surgery in The First Hospital Affiliated to Xiamen University
* Patients with post-operative pathological diagnosis of colorectal cancer

Exclusion Criteria:

* Refuse or fail to cooperate the study (due to any reason)
* Unable to tolerate prehabilitaion strategy (including exercise guide, whey protein and psycho-relaxation exercise)
* Other severe cardio-pulmonary diseases that would affect the 6MWD

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
6-minute-walking-distance (6MWD) | [Time Frame: 4 weeks postoperatively]
  Use 6-minute-walking-distance (6MWD) to evaluate the physical functional capability objectively.

SECONDARY OUTCOMES:
Cancer-related fatigue | [Time Frame: 4 weeks postoperatively]
  Use the Cancer Fatigue Scale to measure the fatigue of cancer patients in the last few weeks,The scale has 3 dimensions, include somatic fatigue, emotional fatigue and cognitive fatigue, with 15 entries. The scale is scored on a 5-point scale. Entries 1, 2, 3, 6, 9, 12, and 15 are used to assess somatic fatigue, 5, 8, 11, and 14 are used to assess emotional fatigue, and 4, 7, 10, and 13 are used to assess cognitive fatigue. The scale has a total score of 0-60, with somatic fatigue scoring in the range of 0-28, emotional fatigue and cognitive fatigue both scoring in the range of 0-16, and the higher the score, the more severe the fatigue.
Quality of Life Scale | [Time Frame: 4 weeks postoperatively]
  Use the SF-36 to evaluate the intermediate phase of recovery.The full scale consists of 25 items, including four dimensions and eight individual items, which are disease information (4 items), medical examination information (3 items), treatment information (6 items), and other service information (6 items). The scale was based on the Likert 4 scale, with answers of "not at all", "somewhat", "quite", and "very "The scores of each dimension/item were linearly converted to a scale of 0-100 according to the EORTC manual, and then the mean value was taken to obtain the total scale score.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Xiamen University, Xiamen, FuJian Provice, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code